CLINICAL TRIAL: NCT02145520
Title: Efficacy of Magnesium Sulfate in the Treatment of Bronchiolitis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12216/12; 12216/12 (Other: Hamad Medical Corporation)
Record Dates: First submitted 2014-01-28; First posted 2014-05-23 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2015-03

CONDITIONS: Bronchiolitis; Magnesium, Abnormal Blood Level
Keywords: bronchiolitis
MeSH Terms: conditions — Bronchiolitis | interventions — Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Magnesium sulfate (Experimental): Magnesium sulfate. Single dose intravenous over one hour.
  Interventions: Drug: Magnesium Sulfate
- placebo (Placebo Comparator): Treatment will be delivered to enrolled patients as currently practice in PEC (Epinephrine nebulization +5%hypertonic saline with/without dexamethasone).
  •All patients will be randomized to receive either Magnesium sulfate over 1 hour or placebo.•Bronchiolitis severity score (BSS) will be recorded at 0, 4, 8, 12, 16,20,24,36,48,60,72 hours, and on discharge.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Magnesium Sulfate — The use of magnesium sulfate intravenous in patient with bronchiolitis in pediatric emergency; follow Broncholitis severity score and length of stay
  Arms: Magnesium sulfate
Other: placebo — use of placebo with standard therapy
  Other Names: normal saline for intravenous.
  Arms: placebo

SUMMARY:
In this study, investigators will compare the efficacy and safety of intravenous (IV) Magnesium sulfate in decreasing bronchiolitis clinical severity score and the duration of hospitalization in admitted patients, as compared to placebo.

DETAILED DESCRIPTION:
* On arrival to Pediatric Emergency Center, patients will be attended by a pediatric specialist on call who will take history and perform full physical examination. Patients will be assessed for eligibility to the study based on the inclusion criteria.
* Guardians of eligible patients will be approached with the study design, objectives and risks; Patients will be included after obtaining a verbal and assigned written consent.
* A chest radiograph and Magnesium level in serum will be requested for all study patients upon recruitment.
* The observation physician will complete the data collection sheet that will include the patient's demographics, physical examination, bronchiolitis clinical severity score,oxygen saturation, chest radiograph findings and Magnesium level.
* Treatment will be delivered to enrolled patients as currently practice in PEC(Nebulized epinephrine 1:1000 1ml in 5 ml of 5% hypertonic saline, every 4 hours until discharge, for all patients and if there is history of Bronchial Asthma in mother, father or full sibling. And/or history of Eczema in the Child ,patients will start on dexamethasone 1mg/kg orally stat.(max-10 mg/dose). Then 0,6 mg/kg orally once daily starting from second day of admission for 4 days).
* All patients will be randomized to receive either Magnesium sulfate intravenous single dose over 1 hour or placebo. And it will be given in the same time with currently practice treatment
* Epinephrine nebulization can be given on PRN basis up to a maximum of every one hour, at a dose of 0.5 mg/kg (min 2.5mg/dose and max 5 mg/dose) mixed in 5 ml of 5% hypertonic saline.•
* Bronchiolitis severity score (BSS) will be recorded at 0, 4, 8, 12, 16,20,24,36,48,60,72 hours, and on discharge.
* Vital signs will be recorded at 0, 2, 4 hours and then every 4 hours from the administration of study medication.
* All patients will be followed up for two weeks post discharge by a phone call asking about the general condition, relapse of symptoms, or need for readmission.

ELIGIBILITY:
Inclusion Criteria:

Infants 1-18 months of age presenting to Al Saad Pediatric Emergency Center from October 2012 to May 2015 with diagnosis of Bronchiolitis and bronchiolitis clinical severity score > 4,will be include in the study.

Exclusion Criteria:

* Prematurity (Gestational age 34 weeks or less);
* Previous history of wheezing;
* Use of steroid within 48 hours of presentation;
* CRITICALLY ill patients with one or more of the following:

  1. obtunded consciousness
  2. progressive respiratory failure requiring intensive care unit (PICU) admission;
  3. history of apnea within 24 hours before presentation
  4. oxygen saturation < 85% on room air at the time of recruitment
* History of chronic lung disease;Chronic lung disease of prematurity Cystic fibrosis;
* Congenital heart disease.
* All immunodeficient children: primary or secondary
* Known hypersensitivity to magnesium sulfate.
* Known to have magnesium or calcium metabolism disturbance. (e.g.; vitamin D deficiency, hypoparathyroidism).

Ages: 1 Month to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2012-10; Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Improvement Percentage of Discharge After a Dose of IV Magnesium sulfate | Time to medical readiness for discharge

SECONDARY OUTCOMES:
Improvement of bronchiolitis clinical severity score | 2 Weeks
  1. Need for admission to ICU during the initial visit
  2. Within 2 weeks after discharge:
     1. Need for clinical revisit
     2. Need for infirmary/observation unit admission
     3. Need for ICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Khalid M Al-Ansai, MD, Principal Investigator — HMC; Rafah F Sayyed, MD, Principal Investigator — HMC
Locations (1):
- Pediatric Emergency Center, Al Saad, Doha, Qatar, Qatar

REFERENCES:
- [Derived] Alansari K, Sayyed R, Davidson BL, Al Jawala S, Ghadier M. IV Magnesium Sulfate for Bronchiolitis: A Randomized Trial. Chest. 2017 Jul;152(1):113-119. doi: 10.1016/j.chest.2017.03.002. Epub 2017 Mar 9. PMID 28286262